CLINICAL TRIAL: NCT01195883
Title: Effect of Goal-directed Crystalloid Versus Colloid Administration on Major Postoperative Morbidity
Acronym: C-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-1051
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-07

CONDITIONS: Postoperative Complications
Keywords: IV fluid; recovery; goal directed fluid replacement; improved patient recovery
MeSH Terms: conditions — Postoperative Complications | interventions — Crystalloid Solutions; Ringer's Lactate; Colloids; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crystalloid (Active Comparator): Lactated Ringers solution will be used for fluid replacement.
  Interventions: Drug: Crystalloid
- Colloid (Active Comparator): Low-molecular weight colloid HES 130/0.4 (Voluven) will be used for fluid replacement
  Interventions: Drug: Colloid

INTERVENTIONS:
Drug: Crystalloid — For goal directed volume management we use corrected aortic flow time (FTc) and stroke volume derived from esophageal Doppler as in previous studies. In case of hypovolemia, detected by esophageal Doppler monitoring (CardioQ, Deltex Medical Group PLC, Chichester, UK) according to a previously published algorithm, an additional fluid bolus of 250 ml of LR will be given over a period of 5 minutes.
  Other Names: Ringer's lactate; Lactated Ringer's solution
  Arms: Crystalloid
Drug: Colloid — For goal directed volume management we use corrected aortic flow time (FTc) and stroke volume derived from esophageal Doppler as in previous studies. In case of hypovolemia, detected by esophageal Doppler monitoring (CardioQ, Deltex Medical Group PLC, Chichester, UK) according to a previously published algorithm, an additional fluid bolus of 250 ml of Hydroxyethylstarch 6% 130/0.4 (Voluven®Fresenius-Kabi, Bad Homburg, Germany) will be given over a period of 5 minutes.
  Other Names: Voluven
  Arms: Colloid

SUMMARY:
A trial in which patients having open abdominal surgery are randomized to receive either crystalloids or colloids intraoperatively, guided by esophageal Doppler. The investigators test the primary hypothesis that goal-directed colloid administration during elective abdominal surgery decreases a composite of postoperative complications within 30 days of surgery.

DETAILED DESCRIPTION:
Patients will be given 5-7 ml/kg of crystalloid (lactated Ringer's) in the immediate preoperative period, which will be followed by 4 ml/kg/h crystalloid for maintenance normalized to ideal body weight [Men: Ideal Body Weight (in kilograms) = 52 kg + 1.9 kg for every 2.5 cm over 150 cm; Women: Ideal Body Weight (in kilograms) = 49 kg + 1.7 kg for every 2.5 cm over 150 cm].

They will then be randomly assigned to additional volume replacement, guided by esophageal Doppler, to either lactated Ringer's solution of Voluven starch.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status 1-3
* Body Mass Index < 35
* Moderate risk elective abdominal surgical procedures scheduled to take ≥ two hours done under general anesthesia.

Exclusion Criteria:

* cardiac insufficiency (EF<35%)
* coronary disease with angina (NYHA IV)
* severe chronic obstructive pulmonary disease
* coagulopathies
* symptoms of infection or sepsis
* renal insufficiency (creatinine clearance <30ml/min or renal replacement therapy)
* ASA Physical Status > 3.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1102 (Actual)
Dates: Start 2010-11; Primary Completion 2016-11 (Actual); Study Completion 2017-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kurz, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (2):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Hillcrest Hospital, Mayfield Heights, Ohio
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reiterer C, Kabon B, Taschner A, Zotti O, Kurz A, Fleischmann E. A comparison of intraoperative goal-directed intravenous administration of crystalloid versus colloid solutions on the postoperative maximum N-terminal pro brain natriuretic peptide in patients undergoing moderate- to high-risk noncardiac surgery. BMC Anesthesiol. 2020 Aug 4;20(1):192. doi: 10.1186/s12871-020-01104-9. PMID 32753064

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crystalloid | Colloid
Started | 553 | 549
Completed | 534 | 523
Not Completed | 19 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crystalloid | Colloid | Total
Number analyzed (Participants) | 534 | 523 | 1057
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (16) | 52 (16) | 52 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268 | 242 | 510
  Male | 266 | 281 | 547

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Morbidity (Major Complications)
Description: Any of the following major complications: (1) Cardiac (Acute heart failure/Myocardial infarction/Ventricular arrhythmia); (2) pulmonary (embolism/edema/respiratory failure/pneumonia/pleural effusion); (3) gastrointestinal (bowel and surgical anastomosis stricture or anastomotic leak/internal or external fistulas/peritoneal effusions); (4) Renal (requiring dialysis); (5) Infectious (deep or organ space surgical site infection / sepsis); and (6) Coagulation (bleeding).
Time Frame: Postoperative 30-days
Measure: Count of Participants; unit: Participants
Arm/Group | Crystalloid | Colloid
Number analyzed (Participants) | 534 | 523
Participants | 103 | 91
Statistical Analysis 1: Comparison: Crystalloid vs Colloid; Test type: Superiority; p = 0.51, GEE model; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.65 to 1.23]

2. Secondary Outcome: Number of Participants With Postoperative Morbidity (Minor Complications)
Description: Any of the following minor complications: (1) unplanned ICU admission; (2) unplanned operation; (3) cardiac (ischemia/non-ventricular arrhythmia/hemodynamic disturbances); (4) pulmonary effusion; (5) deep venous thrombosis; (6) gastrointestinal (effusion/gut paralysis); (7) progressive renal insufficiency; (8) infection (superficial/fever/cystitis or urinary tract infection); and (9) transient neurological injury.
Time Frame: Postoperative 30-days
Measure: Count of Participants; unit: Participants
Arm/Group | Crystalloid | Colloid
Number analyzed (Participants) | 463 | 447
Participants | 234 | 214
Statistical Analysis 1: Comparison: Crystalloid vs Colloid; Test type: Superiority; p = 0.42, Chi-squared; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.81 to 1.11]

3. Secondary Outcome: Number of Participants With Postoperative Complications, 30-day Readmission, and 30-day Death
Description: A composite of the primary outcome, and readmission and death.
Time Frame: Postoperative 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Crystalloid | Colloid
Number analyzed (Participants) | 525 | 518
Participants | 143 | 125
Statistical Analysis 1: Comparison: Crystalloid vs Colloid; Test type: Superiority; p = 0.26, Chi-squared; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.72 to 1.09]

4. Secondary Outcome: Number of Participants With Postoperative Acute Kidney Injury
Description: Preoperative-to-postoperative change in AKIN stage
Time Frame: Hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Crystalloid | Colloid
Number analyzed (Participants) | 527 | 521
Participants | 21 | 16
Statistical Analysis 1: Comparison: Crystalloid vs Colloid; Test type: Superiority; p = 0.40, Chi-squared; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.69 to 2.58]

ADVERSE EVENTS:
Time Frame: 30-days postoperative
Description: Adverse Events were monitored/assessed in such a manner that the specific Adverse Event Terms did not be recorded.
Arm/Group | Crystalloid | Colloid
All-Cause Mortality (participants affected / at risk) | 4/534 | 5/523
Serious Adverse Events (participants affected / at risk) | 103/534 | 91/523
Other Adverse Events (participants affected / at risk) | 234/534 | 214/523
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crystalloid (N=534) | Colloid (N=523)
Cardiac (Cardiac disorders) | 8 (8) | 1 (1) — * Acute heart failure * Myocardial infarction * Ventricular arrhythmia
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 17 (17) — * Pulmonary embolism * Pulmonary edema * Respiratory failure * Pneumonia * Pulmonary pleural effusion
Gastrointestinal (Gastrointestinal disorders) | 51 (51) | 41 (41) — * Bowel and surgical anastomosis stricture/obstruction or anastomotic leak * Internal or external fistulas * Peritoneal effusions
Renal (Renal and urinary disorders) | 4 (4) | 2 (2) — - Requiring dialysis
infections (Infections and infestations) | 58 (58) | 59 (59) — * Deep or organ/space surgical site infection * Sepsis
Coagulation (Vascular disorders) | 12 (12) | 16 (16) — Bleeding
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crystalloid (N=534) | Colloid (N=523)
Minor unplanned operation (Surgical and medical procedures) | 23 (23) | 29 (29)
Cardiac (Cardiac disorders) | 46 (46) | 35 (35) — * Ischemia * Non-ventricular Arrhythmia * Hemodynamic disturbances
Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 46 (46) | 38 (38)
Gastrointestinal (Gastrointestinal disorders) | 103 (103) | 75 (75) — * Effusion * Gut paralysis
Infection (Infections and infestations) | 151 (151) | 139 (139) — Infection * Superficial * Fever * Cystitis or urinary tract Infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No